CLINICAL TRIAL: NCT05602415
Title: A Phase II Study of Postoperative Radiotherapy With Tyrosine Kinase Inhibitor (Anlotinib) for Resectable Soft Tissue Sarcoma With High Recurrence Risk
Brief Title: Anlotinib and Radiotherapy in Resectable Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ2019-200
Record Dates: First submitted 2020-01-21; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Soft Tissue Sarcoma; High Risk of Recurrence; Anlotinib; Radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — anlotinib; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery + Dose Reduced Radiotherapy + Anlotinib (Experimental): Surgery would be performed to resect soft tissue sarcoma with as wide margin as possible. Important vessels and nerves should be preserved.
  Postoperative radiotherapy would be performed. Postoperative intensity-modulated RT (IMRT) will be performed (50 Gy in 2.0 Gy per fraction).
  Anlotinib of 12mg will be administered orally, once daily, 2-days on/1-day off, until disease progression according to RECIST 1.1, death, unacceptable toxicity, or withdrawal of consent for any reasons. A cycle was considered to be 3 weeks. Anlotinib should be started 3-4 weeks after surgery, and continued for 3 months (4 cycles).
  Interventions: Drug: Anlotinib; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Anlotinib — Anlotinib of 12mg will be administered orally, once daily, 2-days on/1-day off, until disease progression according to RECIST 1.1, death, unacceptable toxicity, or withdrawal of consent for any reasons. A cycle was considered to be 3 weeks. Anlotinib should be started 3-4 weeks after surgery, and continued for 3 months (4 cycles). The dose could be reduced to 8-10 mg once daily for patients who had grade 3 or 4 treatment-related toxicities, or for patients with intolerable grade 2 toxicity, despite maximum supportive care measures. If dose reduction was necessary, then the dose of anlotinib was reduced to 10 mg once daily. If further dose reduction was necessary, the dosage was reduced to 8 mg once daily. If the dosage of 8 mg once daily was not tolerable, then the patient stopped receiving anlotinib.
  Other Names: AL3818
Radiation: Radiotherapy — Postoperative radiotherapy would be performed. Postoperative intensity-modu¬lated RT (IMRT) will be performed (50 Gy in 2.0 Gy per fraction). No boost dose would be added if the margin was negative, a boost dose of 10-16 Gy would be added if the margin was microscopically positive, and a boost dose of 16-18 would be added if the margin was gross positive.
Procedure: Surgery — Surgery

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of dose reduced postoperative radiotherapy combined with Anlotinib for patients of soft tissue sarcoma

DETAILED DESCRIPTION:
Right now, resection and radiotherapy (RT) is the most effective and recommended treatment for soft tissue sarcoma (STS). Local recurrence rate has significantly reduced since the application of RT. However, RT has brought a lot of complications which had disturbed patients' quality of life. Anlotinib is a novel tyrosine kinase inhibitor targeting multiple factors involving tumor proliferation, vasculature, and tumor microenvironment. Anlotinib inhibits VEGF/VEGFR signaling by selectively targeting VEGFR-2,-3 and FGFR-1,-2,-3,-4 with high affinity. Anlotinib also suppresses the activity of PDGFRα/β, c-Kit, Ret, Aurora-B, c-FMS, and discoidin domain receptor 1 (DDR1), leading to significant inhibition of tumor proliferation. In phase I study, anlotinib showed promising antitumor potential against STS. In a phase II study, anlotinib showed antitumor activity in several STS with well tolerant and manageable adverse effect.

In this clinical study, investigators will explore the efficacy of Anlotinib combined with dose reduced postoperative radiotherapy on recurrence and metastasis control of STS. Patients with STS would receive standard treatment and recommended dose of radiotherapy. In addition, they will receive anotinib from 3 or 4 weeks after surgery, and continue for 3 months. The primary endpoint is Local Recurrence Free Survival (LRFS).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed and histopathologically confirmed as high histologic grade soft-tissue sarcoma, including undifferentiated pleomorphic sarcoma (UPS), liposarcoma(LPS), leiomyosarcoma (LMS), synovial sarcoma (SS), alveolar soft-part sarcoma (ASPS), clear cell sarcoma (CCS).
2. Upper limb (including shoulder), lower limb (including hip) and pelvic soft-tissue sarcoma,
3. Age ≥ 18 years,
4. High risk of local recurrence was defined if the largest diameter of tumor >5cm and had at least one of below characters (1) Tumor border close (<5mm) to vital tissue (vessel and nerve) from diagnostic MRI (2) MRI shows infiltrative tumor grow type ('focal-type' and 'diffuse-type') (3) Positive microscopic margins or macroscopic residual (4) Recurrent tumor form previous treatment High risk of recurrence must be assessed by staff including a surgeon specialized in sarcoma,
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2,
6. Only one lesion, and can be accurately measured at baseline as ≥ 5cm in the longest diameter with magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements according to RECIST 1.1,
7. Adequate hematological, renal, metabolic and hepatic function:

   Haemoglobin ≥ 9 g/dL and no blood transfusions in the 14 days prior to study entry Absolute neutrophil count (ANc) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L Total bilirubin ≤ 1.5 x upper limit of normality (ULN), Alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) ≤ 2.5 x ULN, Serum creatinine ≤ 150 μmol/L or creatinine clearance ≥ 50 mL/min (according to local institution) in case of serum creatinine > 150 μmol/L, TP, INR ≤ 1.5 x ULN
8. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up,
9. Voluntary signed and dated written informed consent prior to any specific procedure,
10. Patients have a life expectancy of more than 2 years with appropriate therapy,
11. All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

1. Any previous treatment, including chemotherapy, radiotherapy and target therapy, within 6 months from the last time prior to study treatment,
2. Soft-tissue sarcoma occurred at head and neck, visceral organs, retroperitoneum, peritoneum, pelvis within the confines of the bony pelvis
3. Patients with the following entities were excluded: GIST, rhabdomyosarcoma, chondrosarcoma, osteosarcoma, dermatofibrosarcoma protuberans, Ewing sarcoma, primitive neuroectodermal tumor, inflammatory myofibroblastic tumor, and malignant mesothelioma.
4. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication,
5. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy,
6. Patients with known active hepatic disease (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids,
7. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent,
8. Patients with uncontrolled seizures,
9. Women of childbearing potential who are not using an effective method of contraception; women who are pregnant or breast feeding,
10. No prior or concurrent malignant disease diagnosed or treated in the last 2 years,
11. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome,
12. Blood transfusions within 14 days prior to study start,
13. Patients with myelodysplastic syndrome/acute myeloid leukaemia,
14. Major surgery within 6 months of starting study treatment and patients must have recovered from any effects of any major surgery,
15. Participation to a study involving a medical or therapeutic intervention in the last 3 months,
16. Patient unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons,
17. Previous enrollment in the present study,
18. Patients with a known hypersensitivity to study medicines or any of the excipients of the product,
19. Patients with metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Local Recurrence Free Survival (LRFS) | 36-month
  From the time of surgery to the time of local recurrence identified by image examination.

SECONDARY OUTCOMES:
Metastasis free survival (MFS) | 36-month
  From the time of surgery to the time of metastasis identified by image examination.
Overall Survival (OS) | 36-month
  From the time of surgery to the time of death.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | an average of 3 years
  The occurrence of each adverse events(AEs), severe AEs(SAEs) and death according the CTCAE_5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yuhui Shen, MD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China